CLINICAL TRIAL: NCT03913663
Title: A Model Based Study for Gait in Heminglect Patient Pre and Post Vestibul-ocular Rehabilitation
Brief Title: Microsoft Kinect, Gait Function,Hemineglect, Vestibulo-ocular Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mohammed Youssef Elhamrawy, dr, Beni-Suef University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: microsoft kinect hemineglect
Record Dates: First submitted 2019-04-09; First posted 2019-04-12 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-05

CONDITIONS: Hemiplegic Gait
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Active Comparator): 20 patient with hemineglect, minimum 6 months post stroke
  Interventions: Other: vestibuloocular training; Other: regular exercise training for hemiplegic patients
- control group (Active Comparator): 20 patient with hemineglect, minimum 6 months post stroke
  Interventions: Other: regular exercise training for hemiplegic patients

INTERVENTIONS:
Other: vestibuloocular training — using vestibulo ocular training program for training neglect patient
  Other Names: regular exercise training for hemiplegic patients
  Arms: study group
Other: regular exercise training for hemiplegic patients — Traditional gait training program.

SUMMARY:
Gait problems in hemineglect patient post stroke , vestibuloocular training plays a role in improving gait function, gait assessment using a model based study (Microsoft Kinect) for pre and post training assesment.

DETAILED DESCRIPTION:
The syndrome of visuospatial neglect is a common consequence of unilateral brain injury. It is most often associated with stroke and is more severe and persistent following right hemisphere damage, with reported frequencies in the acute stage of up to 80%. This may result in gait disturbance, high levels of energy expenditure and increase the risk of falls. Vestibuleo-ocular training techniques are aimed at improving or even restoring visual function by training patients to detect stimuli in the blind hemifield and increase their overall sensitivity to them. The investigators propose a model based (Microsoft Kinect), a device can be used for assessment of spatiotemporal gait variables as well as gait kinematics.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age will range from (60-70) years old.
* Patients who had a stroke at least six months prior.
* Patients who had visual field defects post stroke.
* Patients who could walk without caretaker assistance or no severe dyskinesias.
* Adequate hearing (hearing aid if required).
* Patients who had no problem with their state of consciousness and absence of dementia
* Patients who had no orthopedic problems that may affect gait.
* Patients will be chosen in both sexes.
* Clinically and medically stable.

Exclusion Criteria:

Patients who will meet one of the following criteria will be excluded from the study:

* Only one functional eye.
* Neurological problem or any severe co-morbidity likely to affect gait.
* Intact visual field.
* Instability of patient's medical condition.
* Obese ( BMI ≥ 30 Kg∕m2 ).
* Association with another medical problem that can affect patient

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-18 (Actual)

PRIMARY OUTCOMES:
gait changes in hemineglect patient after vestibulo ocular rehabilitation program | baseline
  gait assesment using microsoft kinect for hemineglect patient pre and post vestibulo ocular rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: mohammed elhamrawy, master, Principal Investigator — Beni-Suef University
Locations (1):
- Beni Suef University, Banī Suwayf, Beni Suweif Governorate, Egypt

REFERENCES:
- [Background] Gambi E, Agostinelli A, Belli A, Burattini L, Cippitelli E, Fioretti S, Pierleoni P, Ricciuti M, Sbrollini A, Spinsante S. Heart Rate Detection Using Microsoft Kinect: Validation and Comparison to Wearable Devices. Sensors (Basel). 2017 Aug 2;17(8):1776. doi: 10.3390/s17081776. PMID 28767091
- [Background] Basagni B, De Tanti A, Damora A, Abbruzzese L, Varalta V, Antonucci G, Bickerton WL, Smania N, Mancuso M. The assessment of hemineglect syndrome with cancellation tasks: a comparison between the Bells test and the Apples test. Neurol Sci. 2017 Dec;38(12):2171-2176. doi: 10.1007/s10072-017-3139-7. Epub 2017 Oct 4. PMID 28980076
- [Background] Muntaseer Mahfuz M, Schubert MC, Figtree WVC, Todd CJ, Migliaccio AA. Human Vestibulo-Ocular Reflex Adaptation Training: Time Beats Quantity. J Assoc Res Otolaryngol. 2018 Dec;19(6):729-739. doi: 10.1007/s10162-018-00689-w. Epub 2018 Sep 24. PMID 30251187